CLINICAL TRIAL: NCT03985813
Title: Screening Wizard, Component 1 of iCHART (Integrated Care to Help At-Risk Teens)-Feasibility/Pilot Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oliver Lindhiem, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY18110137; P50MH115838-02 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Ultimately, this study design was an open trial after unsuccessful attempts to maintain initial recruitment sites in the study.
  This study initially attempted to use a stepped wedge design, which involves the sequential random rollout of an intervention over 2 time periods. Following a baseline period in which no clusters (= practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.
Masking Description: Outcome assessors will be masked to the intervention condition at follow-up assessment timepoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Wizard (Experimental): Youth and parents receiving Screening Wizard will be screened for depression and suicidal risk within their pediatric primary care provider's office. Screening will be analyzed in real-time to produce a decision support tool meant to guide the primary care provider to make a referral that reflects patient clinical needs and patient and parental treatment preferences and perceived barriers to treatment.
  Interventions: Behavioral: Screening Wizard

INTERVENTIONS:
Behavioral: Screening Wizard — Screening Wizard is a decision support tool to guide the primary care provider to make a referral that reflects patient clinical needs and patient and parental treatment preferences and perceived barriers to treatment.

SUMMARY:
Screening Wizard (SW). Primary Care Providers (PCPs) are often uncertain about how to best refer adolescents who screen positive for depression or suicidality. Screen-positive youth who are either not in treatment, or express dissatisfaction with current treatment will be consented by an on-site research assistant (RA). Those parents and patients receiving SW will answer additional questions: adaptive screens developed in a previous NIMH study (MH100155) for suicidal risk, anxiety, and mania; perceived barriers; and preferences about treatment. SW generates recommendations for PCPs reflecting patient clinical needs and preferences.

DETAILED DESCRIPTION:
Screening Wizard will be delivered by Primary Care Providers (PCPs) at well child visits, beginning with screening occurring within the waiting room which will yield decision support guidance delivered and followed by the PCP at that same visit.

This study utilized an open trial design. A stepped wedge design was originally proposed and efforts were made to adhere to this study design, however after a year of low recruitment and resultant recruitment sites pulling out the of the study, the overall study design was changed to an open trial. Additional recruitment sites were onboarded to the study and provided with the intervention arm in order to obtain feasibility data on the intervention components of the study. For reference a stepped wedge design involves the sequential random rollout of an intervention over two time periods. Following a baseline period in which no clusters (=practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.

Hypothesis: The use of Screening Wizard will increase the rate of personalized referrals experts in specialty mental health would provide, compared to Treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 12-26 yo
* Biological or adoptive parent is willing to provide informed consent for teen to participate
* Youth speaks and understands English

Exclusion Criteria:

* Non English speaking
* No parent willing to provide informed consent
* Is currently experiencing acute mania or psychosis, evidence of an intellectual or developmental disorder (IDD), life threatening medical condition that requires immediate treatment, or other cognitive or medical condition preventing youth from understanding study and/or participating.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Lindhiem, PhD, Principal Investigator — University of Pittsburgh; Ana Radovic, MD, Study Director — University of Pittsburgh
Locations (4):
- United States (4):
  - Children's Community Pediatrics (CCP-Bass Wolfson Cranberry) of Children's Hospital of Pittsburgh of UPMC, Cranberry Township, Pennsylvania
  - Children's Hospital of Pittsburgh Department of Neurology, Pittsburgh, Pennsylvania
  - Children's Primary Care Center (PCC) of Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - UPMC Center for Adolescent and Young Adult Health, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies.
  The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication.
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants were enrolled into the TAU arm prior to converting from a stepped wedge design to an open design.
Groups:
- Treatment As Usual (TAU): Youth and parents randomized to TAU will still be approached to take the Screening Wizard questions, but the resulting report will not be relayed to the treating physician. Imminent suicidality will still be addressed per the practices standard of care. In the TAU condition, the list of depression and suicidality items and based on practice preferences, standard of care substance use items, will be printed and handed to the providers. The handout will not include the decision support tool to guide referrals.
Period: Overall Study
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening Wizard | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 26 | 36
  Between 18 and 65 years | 17 | 0 | 17
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 7 | 14 | 21
  Gender: Female | 17 | 12 | 29
  Gender: Male to Female Transgender | 1 | 0 | 1
  Gender: Female to Male Transgender | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 11 | 14
  White | 19 | 13 | 32
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Personalized Referral
Description: The rate of personalized referrals by primary care providers and treatment initiation among adolescents who screen positive for depression or suicidal ideation will be monitored to determine if provider made referral as recommended on intervention report.
  This initial outcome has been modified as a result of the changes in study design.
Time Frame: Baseline (in office) visit
Population: The number analyzed for each row differs from overall number analyzed as each row is broken into subcategories of recommendations. Not all participants received a specific recommendation. TAU results are recommendations that would have been made based on Screening Wizard algorithm.
Measure: Count of Units; unit: Recommendations
Units Other Than Participants: Recommendations
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Number analyzed (Participants) | 27 | 26
Number analyzed (Recommendations) | 33 | 33
Recommendations
  All recommendations combined: Agree with recommendation | 22 | 15
  All recommendations combined: Disagree with recommendation | 11 | 18
  Watchful Waiting recommendation: number analyzed (Recommendations) | 10 | 10
  Watchful Waiting recommendation: Agree with recommendation | 8 | 10
  Watchful Waiting recommendation: Disagree with recommendation | 2 | 0
  Ask parent further questions recommendation: number analyzed (Recommendations) | 1 | 0
  Ask parent further questions recommendation: Agree with recommendation | 1 | 0
  Ask parent further questions recommendation: Disagree with recommendation | 0 | 0
  Conduct a safety plan assessment recommendation: number analyzed (Recommendations) | 5 | 12
  Conduct a safety plan assessment recommendation: Agree with recommendation | 0 | 0
  Conduct a safety plan assessment recommendation: Disagree with recommendation | 5 | 12
  Refer to embedded therapist recommendation: number analyzed (Recommendations) | 3 | 6
  Refer to embedded therapist recommendation: Agree with recommendation | 1 | 2
  Refer to embedded therapist recommendation: Disagree with recommendation | 2 | 4
  Recommend referral to specialty depression clinic to evaluate suicidality: number analyzed (Recommendations) | 1 | 0
  Recommend referral to specialty depression clinic to evaluate suicidality: Agree with recommendation | 1 | 0
  Recommend referral to specialty depression clinic to evaluate suicidality: Disagree with recommendation | 0 | 0
  Substance use referral recommendation: number analyzed (Recommendations) | 1 | 0
  Substance use referral recommendation: Agree with recommendation | 0 | 0
  Substance use referral recommendation: Disagree with recommendation | 1 | 0
  No treatment needed, rescreen if concern for non-disclosure recommendation: number analyzed (Recommendations) | 10 | 3
  No treatment needed, rescreen if concern for non-disclosure recommendation: Agree with recommendation | 10 | 3
  No treatment needed, rescreen if concern for non-disclosure recommendation: Disagree with recommendation | 0 | 0
  Tobacco counseling recommendation: number analyzed (Recommendations) | 1 | 1
  Tobacco counseling recommendation: Agree with recommendation | 0 | 0
  Tobacco counseling recommendation: Disagree with recommendation | 1 | 1
  Refer to severe anxiety clinic recommendation: number analyzed (Recommendations) | 1 | 0
  Refer to severe anxiety clinic recommendation: Agree with recommendation | 1 | 0
  Refer to severe anxiety clinic recommendation: Disagree with recommendation | 0 | 0
  Refer to mania clinic recommendation: number analyzed (Recommendations) | 0 | 1
  Refer to mania clinic recommendation: Agree with recommendation | 0 | 0
  Refer to mania clinic recommendation: Disagree with recommendation | 0 | 1
Statistical Analysis 1: Comparison: Screening Wizard vs Treatment As Usual (TAU); Test type: Superiority; p = 0.083, Chi-squared — Threshold for significance P<0.05

2. Secondary Outcome: Number of Participants Who Utilized the Screening Wizard Application
Description: Use of the technical components of Screening Wizard will be monitored. Utilization will be measured by the number and proportion of adolescents, parents, and providers who have engaged with the application over time.
Time Frame: Baseline (phone) visit
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Number analyzed (Participants) | 27 | 26
Participants | 27 | 26
Statistical Analysis 1: Comparison: Screening Wizard vs Treatment As Usual (TAU); Test type: Superiority; p > 0.99, Chi-squared — Threshold for statistical significance P<0.05

3. Secondary Outcome: Service Use (Number of Participants at Baseline)
Description: The Child and Adolescent Service Assessment (CASA) will collect service utilization of all participants to determine the amount of services accessed in each treatment arm.
Time Frame: At Baseline phone visit
Population: All participants in both arms responded to CASA questions for Baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Number analyzed (Participants) | 27 | 26
Participants
  Use outpatient services | 19 | 6
  Use school services | 14 | 6
  Use ER services | 2 | 2
  Use legal services | 1 | 0
  Use inpatient services | 3 | 1
  Use medications | 15 | 6

4. Secondary Outcome: Service Use (Number of Participants at 4 Week Follow-up)
Description: as for outcome 3
Time Frame: Week 4 follow-up after Baseline
Population: All Screening WIzard intervention participants responded to 4 week CASA assessment and 25/26 Treatment As Usual participants responded to 4 week CASA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Number analyzed (Participants) | 27 | 25
Participants
  Use outpatient services | 14 | 6
  Use school services | 5 | 4
  Use ER services | 0 | 0
  Use legal services | 0 | 0
  Use inpatient services | 0 | 0
  Use medications | 11 | 3

5. Secondary Outcome: Service Use (Number of Participants at 12 Week Follow-up)
Description: as for outcome 3
Time Frame: Week 12 follow up after Baseline
Population: 26/27 Screening Wizard intervention participants completed CASA assessment and all Treatment As Usual participants completed CASA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
Number analyzed (Participants) | 26 | 26
Participants
  Use outpatient services | 13 | 7
  Use school services | 5 | 3
  Use ER services | 0 | 0
  Use legal services | 0 | 1
  Use inpatient services | 0 | 0
  Use medications | 11 | 4

6. Secondary Outcome: Usability & Satisfaction
Description: Satisfaction to Screening Wizard will be assessed through a question developed by investigators to understand experience with the program. The question investigators have adapted from literature reviews on satisfaction is: "If a friend were in need of a mental health referral, would you recommend Screening Wizard to him/her? The response options include: No, definitely not; No, I don't think so; Yes, I think so; Yes, definitely.
Time Frame: At exit interview after Baseline phone visit. The baseline visit occurs 24-48 hours after initial screening and the exit interview call will be made within 1 month following the completion of the baseline phone assessment.
Population: Out of the 27 participants in the Screening Wizard arm, only 22 answered the satisfaction question at the exit interview. No statistical analysis completed because there is no comparison group.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Wizard
Number analyzed (Participants) | 22
Participants
  No, definitely not | 0
  No, I don't think so | 6
  Yes, I think so | 12
  Yes, definitely | 4

7. Secondary Outcome: Usability & Satisfaction
Description: Satisfaction with the technical components of interventions will be assessed through certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ). The PSSUQ is 19 items with response options ranging from 1 to 7 where 1=strongly disagree and 7=strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. Questions from sub-domains were chosen to tailor the questioning to this particular intervention. Another question about the need to learn new things before using the app was asked to be rated on a 1-5 scale, with 1= strongly disagree and 5= strongly agree.
Time Frame: as for outcome 6
Population: Out of the 27 participants in the Screening Wizard arm, only 19 answered the questions regarding satisfaction with technical components at the exit interview. No statistical analysis completed because there is no comparison group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Screening Wizard
Number analyzed (Participants) | 19
score on a scale
  Overall, I am satisfied with how easy it is to use Screening Wizard | 6.2 (1.3)
  The information such as online help, on-screen messages, and other documentation, provided was clear | 6.2 (1)
  I liked interacting with the Screening Wizard app | 5.7 (1.2)
  I needed to learn a lot of things before I could get going with the Screening Wizard | 1.5 (0.7)

8. Secondary Outcome: Cost Analysis: Cost of Screening Wizard Intervention at Baseline
Description: An overall average of the cost of implementing the Screening Wizard intervention (including labor, equipment, supplies, facilitates) will be estimated at Baseline.
Time Frame: At Baseline
Population: All 27 participants enrolled engaged in using Screening Wizard intervention.
Measure: Mean (Full Range); unit: dollars per participant
Arm/Group | Screening Wizard
Number analyzed (Participants) | 27
dollars per participant | 160.34 [81.54 to 198.88]

ADVERSE EVENTS:
Time Frame: Over the 1 year and 1 month of data collection for the study, participants were assessed for adverse events at each timepoint (baseline, 4 week follow-up, 12 week follow-up)
Arm/Group | Screening Wizard | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

LIMITATIONS AND CAVEATS:
The study design changed from a stepped wedge design to an open trial. As a feasibility trial, the study was not adequately powered to detect significant effects. In some cases, minor issues with the SW decision tree algorithm led to providers in the SW arm receiving guidance for a higher level of care than was necessary. It's possible that some documentation reviewed in the EHR was missing during the consensus and matching process between the EHR referral data and the SW report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03985813/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03985813/ICF_001.pdf